CLINICAL TRIAL: NCT06925828
Title: Application of in Vivo Splitting Technique of Brain-dead Donor Liver in Adult Liver Transplantation
Brief Title: Application of in Vivo Splitting Technique in Adult Liver Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Principal Investigator, lucaide, Professor, Ningbo Medical Center Lihuili Hospital
Other Study IDs: CT2025-LHL-OBS1
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Liver Transplantation
Keywords: Split liver transplantation; Whole liver transplantation; Short-term Outcomes; Surgical complications; Morbidity and Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SLT group: Adult recipients who underwent split liver transplantation
  Interventions: Other: No intervention
- WLT group: Adult recipients who underwent whole liver transplantation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The feasibility of split liver transplantation (SLT) remains controversial. This study aimed to evaluate the outcomes of SLT in adult recipients and to identify specific areas of improvements. A retrospective analysis was conducted on adults who underwent full size SLT between January 2021 and December 2023. The short-term outcomes of these patients who underwent SLT were compared with those of patients who underwent whole liver transplantation (WLT) during the same period.

ELIGIBILITY:
Inclusion Criteria:

* For the donor graft:

  1. age of 18-60 years;
  2. BMI of 19-28 kg/m2;
  3. hemodynamic stability or use of a single vasoactive drug with a small dosage (norepinephrine ≤ 0.1 μg/kg/min or dopamine ≤ 5 μg/kg/min);
  4. liver steatosis ≤ 10%;
  5. liver functional indicators (ALT, AST, total bilirubin quantification) ≤ 3 times the normal value;
  6. blood sodium ≤ 160 mmol/L;

For the SLT recipients

1. Patients who had registered in the China Organ Transplant Response Systems.
2. Initial liver transplantation.
3. Graft-to-Recipient Weight Ratio (GRWR) ≥ 1%.

Exclusion Criteria:

* For the donor graft

  1. uncontrollable infection
  2. significant vascular and biliary variation.

For the recipients

1. Severe portal hypertension.
2. Significant vascular variation.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult recipients who underwent SLT or WLT
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2021.01.01-2025.12.31
  the overall survival of liver transplant recipient during study period

SECONDARY OUTCOMES:
Postoperative complications | 2021.01.01-2025.12.31
  Postoperative complications of liver transplant recipient during study period

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Medical Centre Lihuili Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No